CLINICAL TRIAL: NCT02574650
Title: Early Feasibility of the Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) for Symptomatic Chronic Functional Tricuspid Regurgitation
Brief Title: Early Feasibility of the Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) Also Known as TriAlign™.
Acronym: SCOUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mitralign, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLPR-010
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Chronic Symptomatic Functional Tricuspid Regurgitation; Tricuspid Valve Insufficiency; Heart Valve Disease
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): Non-randomized, open label clinical study that intends to treat up to 30 subjects with the Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) using standard of care techniques and services that are typically used for structural heart procedures.
  Interventions: Device: Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS)

INTERVENTIONS:
Device: Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) — Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) delivered by a percutaneous transcatheter procedure.

SUMMARY:
The purpose of this study is to assess the early safety and performance of the Mitralign Percutaneous Tricuspid Valve Annuloplasty System (PTVAS) for the treatment of symptomatic chronic functional tricuspid regurgitation (FTR).

The procedure will be performed with the PTVAS device using a non-surgical percutaneous approach to tricuspid valve repair in patients who have FTR with a minimum of moderate tricuspid regurgitation.

DETAILED DESCRIPTION:
A prospective, single-arm, multi-center study, enrolling symptomatic patients with chronic functional tricuspid regurgitation and whom left-sided valve surgery is not planned. The study will include up to 30 subjects from up to 6 sites. Follow-up evaluations will be conducted through 2-years post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic functional tricuspid regurgitation (FTR) with a minimum of moderate tricuspid regurgitation;
* ≥18 and ≤85 years old;
* NYHA II - IV;
* Symptomatic despite Guideline Directed medical Therapy (GDMT), at minimum, patient on diuretic use;
* LVEF ≥35%
* Tricuspid valve annular diameter ≥ 40 mm (or 21 mm/m2 (Superscript)) and ≤55 mm (or 29 mm/m2 (Superscript))

Exclusion Criteria:

* Pregnant or lactating female;
* Severe uncontrolled hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg);
* Previous tricuspid valve repair or replacement;
* Severe coronary artery disease;
* MI or known unstable angina within the 30-days prior to the index procedure;
* Any PCI within 30 days prior to the index procedure or planned 3 months post the index procedure;
* Chronic oral steroid use (≥6 months);
* Life expectancy of less than 12-months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Technical success at 30-days | 30-days
  Technical success is defined as freedom from death with: successful access, delivery and retrieval of the device delivery system, and deployment and correct positioning of the intended device(s), and no need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure.

SECONDARY OUTCOMES:
Secondary safety and performance endpoints mid-term and long-term | 24-months with endpoints measured at dishcarge, 1, 3, 6, 12 and 24 months
  The secondary objectives of the study are to evaluate the acute, mid-term and long-term safety of the device and effects of the device on performance, functional and quality of life parameters, as well as technical, procedural and individual patient successes.
Number of participants with a change in Minnesota Living with Heart Failure (MLWHF) Questionnaire and 6-minute walk test (6MWT) as compared to pre-treatment questionnaire responses and pre-treatment total distance walked | 24-months with endpoints measured at dishcarge, 1, 3, 6, 12 and 24 months
  Participants will complete a MLWHF questionnaire and 6MWT before treatment and at each post treatment follow-up check. Percent change over baseline will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hahn, MD, Principal Investigator — Columbia Unviersity Medical Center / New York-Presbyterian Hospital; Christopher Meduri, MD, MPH, Principal Investigator — Piedmont Healthcare
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente, San Francisco, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Delray Medical Center, Delray Beach, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Northwestern University / Bluhm Cardiovascular Institute, Chicago, Illinois
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Columbia University Medical Center / New York-Presbyterian Hospital, New York, New York
  - Houston Methodist, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hahn RT, Meduri CU, Davidson CJ, Lim S, Nazif TM, Ricciardi MJ, Rajagopal V, Ailawadi G, Vannan MA, Thomas JD, Fowler D, Rich S, Martin R, Ong G, Groothuis A, Kodali S. Early Feasibility Study of a Transcatheter Tricuspid Valve Annuloplasty: SCOUT Trial 30-Day Results. J Am Coll Cardiol. 2017 Apr 11;69(14):1795-1806. doi: 10.1016/j.jacc.2017.01.054. PMID 28385308